CLINICAL TRIAL: NCT06392178
Title: SugarVita: an Educative Digital Board Game for Self-management in Diabetes
Brief Title: SugarVita: a Digital Board Game
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Maxima Medical Center (Other)
Responsible Party: Principal Investigator, Edouard Reinders, Principal investigator, Maxima Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: N24.020.
Record Dates: First submitted 2024-04-10; First posted 2024-04-30 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: gamification; mHealth; self-management; diabetes type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SugarVita (Experimental): Participants in the intervention group will download and play the app SugarVita on their mobile phone or tablet, or they can borrow a tablet from the research group. All participants are requested to fill in questionnaires concerning diabetes related topics at the start of the study, and after 8 weeks
  Interventions: Device: SugarVita
- Standard care (No Intervention): Participants in the control group will receive standard care, the usual care that is being given at the outpatient clinic. All participants are requested to fill in questionnaires concerning diabetes related topics at the start of the study, and after 8 weeks

INTERVENTIONS:
Device: SugarVita — Serious digital game (application) that can be played on mobile phone, tablet or personal computer. Self-developed game.
  Arms: SugarVita

SUMMARY:
The serious digital game, SugarVita, is a collaborative effort between the Máxima Medical Centre (MMC) and Eindhoven University of Technology (TUe), intending to enhance self-management for individuals with diabetes. As a mobile application available on smartphones and tablets, SugarVita emerged from cooperative design sessions involving patients diagnosed with diabetes. The average age of type 2 diabetes patients in the Netherlands exceeds 50 years. Following extensive discussions with these patients, the decision was made to model SugarVita after a digital board game, reminiscent of the classic board game 'ganzenbord' (Game of the Goose). In SugarVita, players experience a day in the life of an individual with diabetes, making choices regarding dietary habits, physical activity, and medication intake. Throughout this simulated day, the blood glucose level serves as a central theme. Players earn points by effectively managing their blood glucose levels. SugarVita can be played together with relatives or friends. The game aims to give people with diabetes more control over their chronic condition. Self-care is now seen as the primary approach to diabetes, which is a complex multi-faceted task where training and education are crucial. Importantly, SugarVita recognizes that a conventional 'dry' explanation may not resonate with everyone.

DETAILED DESCRIPTION:
The majority of diabetes mellitus patients in the Netherlands are aged 50 and above, predominantly diagnosed with type 2 diabetes mellitus. Patient education in this context primarily occurs through consultations with healthcare professionals such as general practitioners, internists, and diabetes nurses. However, these interactions alone may not comprehensively address the complexities associated with managing a chronic condition like diabetes. Consequently, self-education constitutes a crucial role in empowering patients to cope with their disease. In response to this need, the investigators have developed SugarVita, a serious game designed to facilitate patient training and skill development in diabetes regulation within the comfort of their homes through playful learning.

Previous studies have indicated that serious diabetes games can enhance patient self-management, potentially leading to controlled or reduced healthcare costs, although the impact on HbA1c levels is often modest. SugarVita distinguishes itself by visualizing the short-term effects of a player's decisions on their glycemic levels and providing rewards for healthy and appropriate choices. The ultimate goal is to encourage the cultivation of health-promoting behaviors in daily life.

SugarVita adopts the format of a digital board game, akin to the Game of the Goose, where players progress through the board by rolling a dice. The SugarVita board comprises a circular arrangement of tiles, mirroring a full day (24 hours), with each tile representing a 20-minute interval. Players traverse the day, encountering various events such as meals, activities, and emotional experiences, all presented in a digital gaming format. The board features distinct pathways corresponding to workdays, outdoor days, and leisure days. Players enter the game through a personalized setup facilitated by the simulator. The primary objective for players is to maintain their glucose levels within a safe range, and therefore earn points by doing so. While immersed in the game, players assume the perspective of an individual with diabetes, navigating the daily decisions inherent to the condition. In this interactive experience, players make choices regarding their food intake, engage in physical activities, and manage medication usage, including insulin doses. The repercussions of these decisions are reflected in the game through a visible glucose meter, dynamically responding to the player's actions. Points are awarded when the glucose meter remains within the target range, creating a learning environment through gameplay and direct feedback. The player achieving the highest score emerges as the winner.

The multiplayer aspect of SugarVita allows patients with diabetes to engage in the game alongside their relatives, fostering discussions about the diverse choices made during gameplay. This collaborative approach enhances mutual understanding of a relative's condition, providing additional support. The unique multiplayer feature of SugarVita distinguishes it from other diabetes games. Involving the social network of patients can potentially contribute to the development of healthier habits.

Designed for the largest segment of diabetes patients, namely young seniors aged 50 to 75 with type 2 diabetes, SugarVita targets lifestyle and habit changes crucial for disease management. Our clinical experience underscores the challenges these patients face in altering their habits and understanding the intricacies of glucose level regulation. Within the young senior demographic, considerable variations exist, including differences in educational attainment and attitudes towards personal health. Some individuals may be illiterate and display minimal concern for their health, while others are motivated to initiate positive changes. Recognizing these differences, the investigators adopted varied approaches to appeal to distinct patient types. Target group interviews further revealed that our audience enjoys board games, expresses openness to digital games, and prefers playing on tablets or mobile phones. While our primary focus is on young senior type 2 patients, SugarVita aims to be appealing to a broader audience, including other diabetes patients, their relatives, and caregivers.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained before trial related activities
* Diagnosed with T2DM
* HbA1c levels > 64 mmol/mol (before start of study)
* BMI > 25 kg/m2
* Age above 18 years
* Patient's language skills are sufficient for participation
* Subject has a smartphone or tablet and is willing to install the needed application on it

Exclusion Criteria:

* Pregnancy or breastfeeding women
* Malignancy except basal and squamous cell skin cancer

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
To assess the impact of SugarVita on self-management | 8 weeks
  This will be measured by filling in the Diabetes Management Self-Efficacy Scale (DSMES) at the beginning of the study (week 1) and at the end (week 8). This is a dutch validated questionnaire consisting of 20 questions. A higher score indicates a higher estimated level of self-management.
To assess the impact of SugarVita on self-confidence | 8 weeks
  This will be measured by filling in the 'Confidence in Diabetes Self-car Scale' questionnaire at the beginning of the study (week 1) and at the end (week 8). This is a dutch validated questionnaire consisting of 20 questions. A higher score indicates a higher estimated level of self-confidence.
To assess the impact of SugarVita on diabetes related knowledge | 8 weeks
  This will be measured by filling in a self created dutch questionnaire concerning questions about diabetes knowledge. This questionnaire will be filled in at the beginning of the study (week 1) and at the end (week 8). This self-developed questionnaire consisting of 19 questions. A higher score indicates a higher estimated level of diabetes related knowledge.

SECONDARY OUTCOMES:
To evaluate the patients perception on SugarVita and the usage of using digital games as an educational tool | 8 weeks
  This will be assed by a self-made questionnaire concerning 11 questions. Participants in the SugarVita group will fill in this questionnaire at the end of the study. Participants in the regular care group do not fill in this questionnaire.
To gather data from player performances in SugarVita (how long do participants play SugarVita in minutes) | 8 weeks
  This data will be collected automatically if participants log into their SugarVita account
To gather data from player performances in SugarVita (how many times do they log into the game, frequency will be measured) | 8 weeks
  This data will be collected automatically if participants log into their SugarVita account

CONTACTS AND LOCATIONS:
Locations (1):
- Maxima Medical Centre, Eindhoven, North Brabant, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided